CLINICAL TRIAL: NCT05681611
Title: Correlation Between Trend of Four Values and Bispectral Index Values During General Anaesthesia for Breast Surgery.
Brief Title: Effect of Rocuronium on BIS Values
Status: Completed | Type: Observational
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Federico Linassi, MD. Anaesthesiologist at Treviso Regional Hospital, University of Padova
Other Study IDs: RocuMAST
Record Dates: First submitted 2022-11-24; First posted 2023-01-12 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer; General Anaesthesia
MeSH Terms: conditions — Breast Neoplasms | interventions — Rocuronium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Rocuronium — Rocuronium bolus was administered, according to our protocol, to facilitate surgery and ventilation.

SUMMARY:
Aim of this trial is to define if Trend of Four (TOF) values after a bolus of rocuronium is correlated with Bispectral Index BIS values during standard general anaesthesia for breast surgery.

DETAILED DESCRIPTION:
Rocuronium. a curarizing agent, has been shown to decrease Bispectral Index (BIS) in awake volunteers.

However, correlation between Trend of Four (TOF) values after a bolus of rocuronium and BIS values during general anaesthesia for breast surgery has not been defined yet.

Investigators want to analyze this correlation during general anaesthesia conducted using Propofol and remifentanil. All of these drugs will be delivered with Targeted-Controlled Infusion pumps (in particular Eleveld for Propofol, Minto for Remifentanil), commonly used to deliver general anaesthesia. At stable anaesthesia maintenance, if requested for surgical (ie more muscle relaxation) or anesthesiological reasons (i.e. avoid air insufflation) a standard Rocuronium bolus (0.6 mg/kg) was given. In these case, with rocuronium bolus justified by clinical reasons, authors will observationally record the BIS values and the TOF values.

ELIGIBILITY:
Inclusion Criteria:

* Undergo General Anaesthesia with Propofol and Remifentanil, and necessity of curarization with Rocuronium for surgical or ventilatory reasons.

Exclusion Criteria:

* Neurological disease
* Psychiatric disease
* Benzodiazepines praemedication
* Obesity

Ages: 18 Years to 80 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Fe-male patients undergoing breast oncologic surgery
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2023-03-03 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Correlation between Trend of Four (TOF) and Bispectral Index (BIS) values | 60 minutes after rocuronium bolus
  Discover if there is linear correlation between TOF values (utilized for curarization monitoring) and BIS values (utilized for deep of hypnosis monitoring) during standard general anaesthesia conducted with Propofol and remifentanil with targeted controlled infusion pumps, usually adopted in our Hospital to delivery general anaesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- ULSS2, Treviso, Italy

IPD SHARING:
Plan to Share IPD: Undecided